CLINICAL TRIAL: NCT02733367
Title: Open-label, Long-term Follow-up of Safety and Biochemical Disease Control of Infacort® in Neonates, Infants and Children With Congenital Adrenal Hyperplasia and Adrenal Insufficiency Previously Enrolled in the Infacort 003 Study
Brief Title: Extension Study for Patients Entered Into Study Infacort 003
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Infacort 004
Record Dates: First submitted 2016-03-16; First posted 2016-04-11 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infacort (Experimental): Infacort® granules
  Interventions: Drug: Infacort®

INTERVENTIONS:
Drug: Infacort® — Infacort® is a dry granule formulation of hydrocortisone stored in capsules available in different strengths (0.5, 1.0, 2.0 and 5.0 mg).

SUMMARY:
A Phase 3, open-label, single-group, non-randomised, observational study of the safety and biochemical disease control of Infacort® in neonates, infants and children with adrenal insufficiency and congenital adrenal hyperplasia who had completed study Infacort 003. All subjects who had satisfactorily completed study Infacort 003 were offered the opportunity to take part in Infacort 004.

DETAILED DESCRIPTION:
A Phase 3, open-label, single-group, non-randomised, observational study of the safety and biochemical disease control of Infacort® in neonates, infants and children with AI who had completed study Infacort 003 (EudraCT number 2014-002265-30). All subjects who had satisfactorily completed study Infacort 003 wiere offered the opportunity to participate in study Infacort 004 at or after their final visit of study Infacort 003. Subjects received the usual clinically-appropriate dose (since bioequivalence has been demonstrated with conventional hydrocortisone), as determined by the Investigator, which was administered according to usual clinical practice - generally 3 or 4 times a day. Subjects could continue to be treated in this study until they met the study withdrawal criteria, until Infacort® was commercially available locally (which has now been achieved), or until the Sponsor decided to discontinue the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects successfully completing study Infacort 003, whose inclusion criteria were:

1. Male and female children less than 6 years of age.
2. A diagnosis of adrenal insufficiency (AI) as confirmed by an inappropriately low cortisol usually with other supporting tests.
3. Receiving appropriate adrenocortical replacement therapy (hydrocortisone with/without fludrocortisone).
4. Adequately hydrated and nourished. In addition, the parents/carers must be able to understand and give written Informed Consent for this extension study.

Exclusion Criteria:

1. Clinically evident acute AI (adrenal crisis) (Note: the subject can be re-evaluated for eligibility once the episode is over)
2. Inability of the child to take oral therapy
3. Subjects with clinical signs of acute infection or fever on inclusion (Note: the subject can be re-evaluated for eligibility once the episode is over)
4. Any surgical or medical condition that in the opinion of the Investigator may place the subject at higher risk from his/her participation in the study
5. Parents/carers of subjects unwilling to consent to saving and propagation of pseudonymised medical data for study reasons
6. Subjects who are in a dependent relationship with the Investigator or the Sponsor

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wiegand, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Universitätsmedizin Berlin, CVK, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Infacort: Infacort® granules
  Infacort®: Infacort® is a dry granule formulation of hydrocortisone stored in capsules available in different strengths (0.5, 1.0, 2.0 and 5.0 mg). This was a non-randomised, open-label, single-group study; all subjects who participated received Infacort. One subject was initially withdrawn from the study, but subsequently re-enrolled.
Period: Overall Study
Arm/Group | Infacort
Started | 18
Completed | 12
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Subjects recruited were those who had satisfactorily completed study Infacort 003 and agreed to participate in study Infacort 004. The investigator ensured that all subjects who were treated in study Infacort 003 were invited to participate.
Arm/Group | Infacort
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 1021.6 (650.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 18
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 17.02 (2.083)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 0.582 (0.1803)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: The primary endpoint was the nature and occurrence of serious adverse events (SAEs) and adverse events (AEs) observed throughout the study. AEs were recorded from the time of the first intake of Infacort until the final visit.
Time Frame: 29 months
Measure: Number; unit: adverse events
Arm/Group | Infacort
Number analyzed (Participants) | 18
adverse events
  Treatment-Emergent Adverse Events (TEAE) - Overall | 193
  Serious TEAEs | 9
  Severe TEAEs | 0
  Moderate TEAEs | 42
  Mild TEAEs | 151

2. Secondary Outcome: Growth Velocity
Description: Growth velocity standard deviation score (SDS). Body height/length (cm) was obtained at each visit by specially trained paediatric endocrine nurses or physicians using standard calibrated auxological methods.
Time Frame: 29 months
Population: Reference data for growth velocity is only available for patients <=6 years old at time of assessment. Therefore n=2 & not 4 for C1 at Month 11. Subject 001 was re-enrolled so no Visit 10 data available and, therefore, n=1 for C1 at Month 23.
Measure: Mean (Standard Deviation); unit: Standard Deviation Score
Arm/Group | Infacort
Number analyzed (Participants) | 10
Standard Deviation Score
  visit 6 - 11th Month | 0.6343 (2.51996)
  Visit 10 - 23rd Month: number analyzed (Participants) | 9
  Visit 10 - 23rd Month | 0.9214 (1.88757)

3. Secondary Outcome: Cortisol Levels
Description: Cortisol levels measured from dried blood spots. The dried blood spots were analysed for multi-steroids, including cortisol (all subjects). Blood spot absolute laboratory values for the safety population are presented. A dried blood spot sample was collected at the initial and final visits, every month for the first 2 months of the study and thereafter every 6 months (unless required after 3 months).
Time Frame: 29 months
Population: The reason why n=14 at Visit 1 is because of no result for Subjects 005, 010, 017 & 018. N=12 at Final Visit due to 12 completers.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Infacort
Number analyzed (Participants) | 17
nmol/L
  Visit 1: number analyzed (Participants) | 14
  Visit 1 | 43.329 (48.3217)
  Final Visit: number analyzed (Participants) | 12
  Final Visit | 22.022 (27.1323)

4. Secondary Outcome: Number of Participants Exhibiting a Change in Tanner Development Stage
Description: The Tanner Development Stage was assessed as an additional analysis in this study. All assessments (breast, genitalia, and pubic hair) were Grade 1 (pre-pubertal) at baseline, with only 1 subject (in Cohort 2) showing a change during the study. Subject 018 showed progression to Grade 2 in the pubic hair category (sparse, pigmented hair mainly on labia).
Time Frame: 29 months
Population: 'Count of Participants' data below represents the number of subjects that exhibited a change from baseline in their Tanner Development Stage.
Measure: Count of Participants; unit: Participants
Arm/Group | Infacort
Number analyzed (Participants) | 18
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of the first intake of Infacort in this study until the final study visit (i.e. 29 months).
Description: Details of any adverse events were collected, including date of onset, end date, frequency, severity, seriousness, relationship to Infacort, action taken, and outcome. Any adverse event was followed, whenever possible, until it returned to the baseline condition or became stable with no further change expected.
Arm/Group | Infacort
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infacort (N=18)
Vomiting (Gastrointestinal disorders) | 1 (2)
Erysipelas (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (4)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infacort (N=18)
Secondary hypertension (Vascular disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Venomous sting (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 1 (1)
Genitourinary operation (Surgical and medical procedures) | 2 (2)
Circumcision (Surgical and medical procedures) | 1 (1)
Body temperature increased (Investigations) | 2 (6)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (3)
Paraesthesia (Nervous system disorders) | 1 (2)
Pyrexia (General disorders) | 10 (45)
Abdominal pain (Gastrointestinal disorders) | 1 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (6)
Nausea (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 6 (12)
Vulval disorder (Reproductive system and breast disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (6)
Conjunctivitis (Infections and infestations) | 5 (6)
Enterovirus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 8 (11)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (2)
Otitis media viral (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 2 (2)
Pharyngotonsilitis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2)
Roseola (Infections and infestations) | 1 (1)
Tonsilitis (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 6 (6)
Viral upper respiratory tract infection (Infections and infestations) | 7 (21)
Scarlet fever (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was designed as a safety study to evaluate the long-term use of Infacort in routine clinical practice. Efficacy results should be viewed as exploratory and interpreted with care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT02733367/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02733367/SAP_001.pdf